CLINICAL TRIAL: NCT02655874
Title: A Single-centre, Randomised, Observer-blind, Active Comparator-controlled, Superiority Trial of the Immune Response to Six-monthly Versus Annual Standard Dose Inactivated Trivalent Influenza Vaccination in the Elderly
Brief Title: Tropical Influenza Control Strategies for the Elderly
Acronym: TROPICS1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: National Healthcare Group, Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015/01047
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Influenza, Human
Keywords: Seasonal Influenza; Antibody response; Influenza Vaccines; Hemagglutination Inhibition; Elderly; immunosenescence; Tropics
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Diphtheria-Tetanus-Pertussis Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Six-monthly influenza vaccine (Experimental): Standard dose trivalent inactivated seasonal influenza vaccine will be administered at day 1 and 180
  Interventions: Biological: Influenza vaccine
- Annual influenza vaccine (Active Comparator): Standard dose trivalent inactivated seasonal influenza vaccine will be administered at day 1 and an active-comparator (Tetanus-diphtheria-pertussis) at day 180
  Interventions: Biological: Influenza vaccine; Biological: Tetanus-diphtheria-pertussis vaccine

INTERVENTIONS:
Biological: Influenza vaccine — Administered at day 1
Biological: Influenza vaccine — Administered at day 180
  Arms: Six-monthly influenza vaccine
Biological: Tetanus-diphtheria-pertussis vaccine — Administered at day 180
  Arms: Annual influenza vaccine

SUMMARY:
TROPICS1 is a randomized, observer-blind, active comparator-controlled, single-center, Phase IV trial in 200 participants aged ≥65 years. The control group will receive a standard dose licensed trivalent inactivated influenza vaccine at day 1, and an active-comparator (Tetanus-diphtheria-pertussis vaccine) at day 180. Participants in the experimental group will receive the same influenza vaccine at day 1 and day 180. Endpoints are immunological, and include measures of haemagglutination-inhibition (HI) titres, micro-neutralisation titres and cell-mediated immunity at 4 time points after the initial vaccination up to Day 360. The primary hypothesis is that participants receiving an influenza booster at day 180 will achieve superior influenza seroprotection (HI titre ≥1:40) at day 208, compared to controls.

The World Health Organization (WHO) estimates the global annual burden from seasonal influenza as 1 billion infections, with 3-5 million severe cases and 300,000-500,000 deaths. The pattern and impact of these infections varies considerably with climate. In temperate countries, influenza epidemics characteristically occur during the cold winter months, while in sub-tropical countries, they coincide with the rainy seasons. Closer to the equator, influenza virus activity is more complex. In Singapore, biannual epidemics are usual, but with continuous transmission year-round. Bi-annual epidemics, tri-annual epidemics and year round virus activity have also been described in other tropical countries, from Indonesia and Malaysia to Peru and Mexico.

There is no published data reporting year-round influenza vaccine effectiveness in the elderly from countries with continuous influenza virus activity. Despite numerous studies worldwide exploring the HI antibody response to influenza vaccination, the majority of these do not continue follow up beyond seroconversion (21-28 days). However, of the few available, HI antibody titres declined following influenza vaccination in the elderly, such that within 6-12 months geometric mean titres approached pre-vaccination levels. With biannual epidemics and year-round transmission in tropical regions, year-round seroprotection may be important to reduce influenza infections in this environment. A six-monthly vaccination cycle would correspond with the decline in vaccine-induced seroprotection in the elderly, and the 6-monthly periodicity of outbreaks in Singapore and other tropical countries.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥65 years on the day of inclusion
2. No influenza vaccination in the previous 10 months
3. No tetanus, diphtheria or pertussis vaccine in the previous 1 year
4. No virologically confirmed influenza infection in the previous 10 months
5. Able to provide written informed consent
6. Able to attend all scheduled visits and comply with all trial procedures

Exclusion Criteria:

1. Participation in the 4 weeks preceding the first trial vaccination or participation during the present trial period in another trial investigating a vaccine, drug, medical device, or medical procedure
2. History of a life threatening reaction to the vaccine used in the trial, or to a vaccine containing any of the same substances
3. Known systemic hypersensitivity to any of the vaccine components, including:

   * Egg protein (eggs or egg products)
   * Chicken products
   * Formaldehyde
   * Neomycin or kanamycin
   * Octoxinol 9 (Triton X-100)
   * Cetyltrimethylammonium bromide (CTAB)
4. History of Guillain-Barré syndrome (GBS) within 6 weeks following previous influenza vaccination
5. Acute respiratory infection on the day of enrolment
6. Moderate or severe acute illness/infection (according to investigator judgement) on the day of vaccination, or febrile illness (temperature ≥ 37.5°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided.
7. Self-reported thrombocytopenia, contraindicating Intramuscular vaccination
8. Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding six months; or long-term systemic corticosteroid therapy (prednisolone ≥ 7.5mg/day or equivalent for more than 2 consecutive weeks within the past 3 months)
9. Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
10. Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
11. Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures in the opinion of the Investigator

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Seroprotection (Proportion of subjects with HI titre ≥1:40 (1/dil) at day 208 post-primary vaccination for each of the influenza strains present in the administered influenza vaccine) | Day 208 post-vaccination
  Proportion of subjects with HI titre ≥1:40 (1/dil) at day 208 post-primary vaccination for each of the influenza strains present in the administered influenza vaccine.

SECONDARY OUTCOMES:
Geometric mean titres | Day 208 to 360 post-vaccination
  Comparison by vaccination group of Geometric mean titres (GMTs) post-primary vaccination against homologous and heterologous influenza strains to those present in the administered influenza vaccine.
Geometric mean ratio | Day 208 to 360 post-vaccination
  Comparison by vaccination group of the Geometric mean ratio (GMR) post-primary vaccination against homologous and heterologous influenza strains to those present in the administered influenza vaccine.
Seroprotection (Proportion of subjects with HI titre ≥1:40 (1/dil) at day 208 post-primary vaccination for each of the influenza strains present in the administered influenza vaccine) | Day 360 post-vaccination
  Comparison by vaccination group of the proportion of subjects with HI titre ≥1:40 (1/dil) at day 360 post-primary vaccination for each of the influenza strains present in the administered influenza vaccine.
Seroconversion (Proportion of subjects achieving seroconversion after vaccination for each of the influenza strains present in the administered influenza vaccine) | Day 208 to 360 post-vaccination
  Comparison by vaccination group of the proportion of subjects achieving seroconversion after vaccination for each of the influenza strains present in the administered influenza vaccine. Seroconversion is defined as a pre-vaccination HI titre < 1:10 and a post vaccination titre ≥1:40, or a pre-vaccination titre > 1:10 and a minimum fourfold rise in HI titre.
Micro-neutralization titres | Day 208 to 360 post-vaccination
  Comparison by vaccination group of Micro-neutralization titres post-primary vaccination against strains present in the administered influenza vaccine.
Influenza-like illness | Day 208 to 360 post-vaccination
  Comparison by vaccination group of the number of subjects reporting an influenza-like illness
Influenza infection | Day 208 to 360 post-vaccination
  Comparison by vaccination group of the number of subjects with PCR confirmed influenza infection
Healthcare utilization | Day 180 to 360 post-vaccination
  Comparison by vaccination group of the number of subjects reporting healthcare utilization. This is defined as unscheduled physician visits, emergency room visits and hospitlizations.
Solicited and unsolicited adverse events | Day 1 to 7 and day 180 to 187
  Frequency and severity of solicited local (injection site) and systemic adverse events for 7 days post-vaccination
Serious adverse events | Day 1 to 28, and day 180 to 208
  A serious adverse event is defined as any untoward medical occurrence that is an important event.

CONTACTS AND LOCATIONS:
Overall Officials: Barnaby Young, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Institute of Infectious Disease and Epidemiology, Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Young B, Sadarangani S, Haur SY, Yung CF, Barr I, Connolly J, Chen M, Wilder-Smith A. Semiannual Versus Annual Influenza Vaccination in Older Adults in the Tropics: An Observer-blind, Active-comparator-controlled, Randomized Superiority Trial. Clin Infect Dis. 2019 Jun 18;69(1):121-129. doi: 10.1093/cid/ciy836. PMID 30277500
- [Derived] Young B, Sadarangani S, Yew HS, Yung CF, Leo YS, Chen MI, Wilder-Smith A. The immune response to 6-monthly versus annual standard dose inactivated trivalent influenza vaccination in older people: study protocol for a randomised clinical trial. Trials. 2017 Feb 10;18(1):67. doi: 10.1186/s13063-017-1808-8. PMID 28183326